CLINICAL TRIAL: NCT06321432
Title: Intensive Weight Loss Intervention Versus Usual Care for Adults With Obesity: the LightCARE Randomised Trial. Lighthouse Consortium on Obesity Management (LightCOM) Trial no 2
Brief Title: Intensive Weight Loss Intervention Versus Usual Care for Adults With Obesity
Acronym: LightCARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carsten Dirksen (Other)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other); University of Oxford (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Carsten Dirksen, Associate Professor, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LightCARE
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the interventions, it will not be possible to blind the participants or the healthcare providers administering the interventions. In all other aspects of the trial, blinding will be employed. Outcome assessors will be blinded to group allocation. Participants will also be requested not to disclose their allocation when outcomes are assessed.
  Statisticians and investigators drawing conclusions will be fully blinded. The statistical analyses will be conducted with the intervention groups coded as e.g., 'A' and 'B'. The Steering Committee ill write two abstracts while the blinding is intact; one assuming the experimental intervention group is 'A' and the control intervention group is 'B', and one assuming the opposite. After these two abstracts have both obtained consensus, the code will be broken by the data manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive weight loss intervention (Experimental): The intensive weight loss intervention (IWL) includes total dietary replacements, behavioural support, and weight loss medication. The intervention consists of three phases: induction, weight loss continuation, maintenance, and it will lasts two years in total.
  Interventions: Behavioral: Intensive weight loss intervention
- Usual care (Active Comparator): Denmark: usual care offered by the GP or local municipality. The UK: usual care in primary care, Tier 2 weight management services.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Intensive weight loss intervention — Intensive weight loss intervention, incl. total meal replacements, behavioural support, and weight loss medication.
  Arms: Intensive weight loss intervention
Behavioral: Usual care — Usual care
  Arms: Usual care

SUMMARY:
In this trial, the aim is to assess the clinical benefits and harms, as well as cost-effectiveness of an intensive weight loss (IWL) intervention that includes total dietary replacements, behavioural support and weight-loss medication compared with existing weight management programmes within primary care for people with obesity class I or uncomplicated obesity class II or higher.

DETAILED DESCRIPTION:
In the LightCARE trial, an intensive weight loss (IWL) intervention will compared with usual care. The IWL lasts two years, and includes total dietary replacements, behavioural support, and weight loss medication in three phases:

* Induction' phase (week 0-12 after randomisation): total dietary replacement (TDR) programme and behavioural support with weight loss medication (WLM) if rate of weight loss is insufficient.
* Weight loss continuation' phase (week 13-32 after randomisation): progression of dietary programme including reduction in use of TDR products, reintroduction of healthy foods, with behavioural support, introduction of physical activity, WLM (as required).
* Maintenance' phase (week 33-104 after randomisation): Continued healthy diet and physical activity with WLM (if required), with return to induction phase if weight regain occurs induction, weight loss continuation, maintenance.

Usual care will differ between the two countries (Denmark and the United Kingdom).

In Denmark, participants will receive a pamphlet on current obesity management guidelines from the Danish National Board of Health, and will be advised to contact their GP for potential referral to local municipality-based obesity management programmes. Furthermore, a notification will be sent to the participant's GP, informing that the participant has been enrolled in the trial and is randomised to usual care. The availability and structure of current obesity programmes varies between municipalities.

In the United Kingdom, participants will be offered to discuss weight management programmes available in their area with their GP practice; the programmes available referral routes vary slightly from place to place. Tier 2 weight management services are mostly commissioned by local authority, and therefore differ slightly across the 333 local authorities in England. These local community-based weight management services provide diet, nutrition, behavioural advice.

ELIGIBILITY:
Please note that participants need to be invited in order to take part in the trial.

Inclusion Criteria:

1. Age ≥18 years and ≤60 years old at screening.
2. BMI ≥30 kg/m2 or ≥27.5 kg/m2 in people with South Asian, Chinese, other Asian, Middle Eastern, Black African or African-Caribbean family backgrounds (as reported by the participants).
3. Informed consent.

Exclusion Criteria:

1. Has severe and complex obesity, i.e., obesity class II (BMI≥35 if white or 32.5 if non-white) with one or more of these specific adiposity-related comorbidities: cardiovascular disease, type 2 diabetes, hypertension, non-alcoholic steatosis, or sleep apnoea (Appendix 1).
2. Intending to become pregnant in the next two years, or pregnant, or breastfeeding.
3. Use of WLM or GLP-1 agonist treatment within the last 3 months.
4. Currently being treated for cancer other than oestrogen antagonist therapy or non-melanoma skin cancer.
5. Prior bariatric surgery, not including laparoscopic gastric banding, intragastric balloons or duodenal-jejunal bypass sleeve (Endobarrier™ or similar) if the device has been removed >1 year before screening.
6. Diagnosis or treatment for eating disorder within the last 6 months.
7. Any other disease that markedly compromises the participant's ability to adhere to the treatment programme or follow-up or is likely to mean that weight loss will not improve the person's length or quality of life, such as conditions limiting life expectancy.
8. Conditions that contraindicate or complicate total diet replacement (including type 1 diabetes or other diabetes requiring any insulin therapy, phenylketonuria, or other conditions requiring special diets).
9. Taking part in other research involving multidisciplinary obesity treatment that would compromise participation in this trial.
10. Conditions that contraindicate or complicate GLP-1 or GIP agonist treatment (including history of pancreatitis)
11. Another member of the household enrolled in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2048-12 (Estimated)

PRIMARY OUTCOMES:
Weight | 104 weeks after randomisation
  Weight (kg)

SECONDARY OUTCOMES:
Weight loss (20%) | 104 weeks after randomisation
  Proportion of participants with weight loss ≥20%
Short-Form-36, mental component score | 104 weeks after randomisation
  Quality of life, SF36-mental component score (scale from 0-100, higher scores indicate better mental health)
Gait speed | 104 weeks after randomisation
  4-metre gait speed (m/s)
MetS-Z | 104 weeks after randomisation
  Metabolic syndrome severity Z-score (scale from -4 to 4, mean is 0, higher scores indicate a worse outcome)

OTHER OUTCOMES:
Safety - SAE | 104 weeks after randomisation
  Proportion of participants that experienced at least one serious adverse event (according to ICH-GCP guidelines)
Safety - eating disorder | 104 weeks after randomisation
  Proportion of participants with incident eating disorders during the intervention period
Safety - bone mineral density (BMD) assessed by DXA | 104 weeks after randomisation
  1. Bone mineral density (g/cm²) of hip (total hip and femoral neck).
  2. Bone mineral density (g/cm²) of lumbar region.
Body composition - waist circumference | 104 weeks after randomisation
  Waist circumference (cm)
Body composition - fat percentage | 104 weeks after randomisation
  * Body fat percentage
  * Visceral fat percentage
  * Subcutaneous fat percentage
Body composition - weight loss (10%) | 104 weeks after randomisation
  Proportion of participants with weight loss ≥10%
Physical functioning - SENS | 104 weeks after randomisation
  Objectively measured moderate to vigorous physical activity (MVPA) using SENS Motion accelerometers (hours/day)
Physical functioning - SF-36 | 104 weeks after randomisation
  Short Form 36 (SF-36) physical component score (scale from 0-100, higher scores indicate better physical health)
Physical functioning - sit to stand test | 104 weeks after randomisation
  Number of sit to stands completed 30 Second Sit to Stand test
Physical functioning - quality of life | 104 weeks after randomisation
  EQ-5D-5L (the 5-level EQ-5D version), index score (score between -1 and 1, higher scores indicate better health)
Sleep | 104 weeks after randomisation
  Sleep duration using SENS Motion accelerometers (hours/day)
Medications during the intervention period | 104 weeks after randomisation
  1. Proportion of participants prescribed glucose-lowering medications during the intervention period (number, type)
  2. Proportion of participants prescribed lipid-lowering medications during the intervention period (number, type)
  3. Proportion of participants prescribed blood pressure-lowering medications during the intervention period (number, type)
  4. Proportion of participants prescribed medication for pain relief during the intervention period (number, type)
  5. Proportion of participants prescribed medications for psychiatric disorders (number, type)
Metabolic health - blood pressure | 104 weeks after randomisation
  Systolic and diastolic blood pressure (mmHg)
Metabolic health - pulse | 104 weeks after randomisation
  Pulse rate (beats per minute)
Metabolic health - glucose | 104 weeks after randomisation
  Fasting glucose concentration (mmol/l)
Metabolic health - Hb1Ac | 104 weeks after randomisation
  Haemoglobin A1c (mmol/mol)
Metabolic health - insulin | 104 weeks after randomisation
  Fasting insulin concentration (pmol/L)
Metabolic health - HOMA2-IR | 104 weeks after randomisation
  HOMA2-IR (calculated from glucose and C-peptide concentration) (ratio)
Metabolic health - lipids | 104 weeks after randomisation
  Fasting lipid profile (HDL, LDL and triglycerides) (mmol/L)
Metabolic health - eGFR | 104 weeks after randomisation
  Estimated Glomerular Filtration Rate (eGFR), creatinine (µmol/L), calculated from creatinine, sex and years
Metabolic health - hsCRP | 104 weeks after randomisation
  High-sensitivity C-reactive protein (hsCRP), mg/L
Metabolic health - Fib4 | 104 weeks after randomisation
  Fib-4 (ALT/AST/platelets) (ratio)
Metabolic health - Proteinuria | 104 weeks after randomisation
  Proteinuria, measured as urine albumin/creatinine (ratio)
Metabolic health - TSH | 104 weeks after randomisation
  Thyroid-stimulating hormone (IU/L)
Mental health - MDI | 104 weeks after randomisation
  Major Depression Inventory (MDI) (scale from 0-50, higher scores indicate more symptoms of depression)
Mental health - WBIS-M | 104 weeks after randomisation
  Weight Bias Internalization Scale (WBIS-M) score (scale from 1-7, higher scores indicate higher degree of internalised weight bias)
Mental health - EDE-Q | 104 weeks after randomisation
  Eating Disorder Examination Questionnaire (EDE-Q) score (scale from 0 to 6, higher scores indicate higher degree of eating disorder)
Labour market attachment - WPAI | 104 weeks after randomisation
  Work productivity and impairment (WPAI) score points (scale from 0-100, higher scores indicate more limitations in ability to work and lower productivity)
Labour market attachment - days of sick leave | 104 weeks after randomisation
  Self-reported number of days sick leave during follow-up
Genetic profiles' (using comprehensive genetic mapping) association with the metabolic and/or weight loss response to IWL vs usual care | 104 weeks after randomisation
  1. Common gene variants with low to moderate effect on the phenotype for the construction of aggregate genetic risk scores
  2. Rare variants with potential functional effects in genes known to harbour high-impact obesity variants e.g. MC4R, LEP, LEPR, POMC, PCSK1, SIM1, NTRK2, MC3R, MRAP2, BDNF, SH2B1, KSR2
Health economy: Within-trial cost-effectiveness analysis - quality of life | 104 weeks after randomisation
  Quality of life (measured using the 5-level EQ-5D version (EQ-5D-5L), VAS score (scale from 0-100, higher scores indicate better health)
Health economy: Within-trial cost-effectiveness analysis - costs | 104 weeks after randomisation
  24-month costs, DKK
Health economy: Within-trial cost-effectiveness analysis - QALY | 104 weeks after randomisation
  Incremental cost per quality-adjusted-life-year (QALY) gained, DKK
Health economy: Model-based cost-effectiveness analysis - QALY | 104 weeks after randomisation
  Predicted lifetime QALYs gained
Health economy: Model-based cost-effectiveness analysis - healthcare costs | 104 weeks after randomisation
  Predicted lifetime healthcare costs, DKK
Health economy: Model-based cost-effectiveness analysis - cost effectiveness ratios | 104 weeks after randomisation
  Long-term incremental cost effectiveness ratios
Long-term effects - mortality and major cardiovascular disease (CVD) | 5, 10 and 20 years after randomisation
  * Proportion of participants who die from any cause
  * Proportion of participants with a major CVD outcome consisting of any of the following (each of the components will be assessed exploratively): myocardial infarction, stroke, hospitalisation for angina, coronary-artery bypass grafting, percutaneous coronary intervention, hospitalisation for heart failure, peripheral vascular disease
Long-term effects - prescription patterns | 5, 10 and 20 years after randomisation
  1. Proportion of participants on glucose-lowering medications
  2. Proportion of participants on lipid-lowering medications
  3. Proportion of participants on blood pressure-lowering medications
  4. Proportion of participants on medication for pain relief
  5. Proportion of participants on weight loss medication
  6. Proportion of participants on medication used for psychiatric disorders (antidepressants, anxiolytics, antipsychotics)
Long-term effects - incident cancer | 5, 10 and 20 years after randomisation
  1. Proportion of participants with any diagnosis of cancer
  2. Proportion of participants with cancers known to be associated with obesity: GI tract including liver and kidney and reproduction organs (including breast for women and prostate for men)
Long-term effects - fracture risk | 5, 10 and 20 years after randomisation
  1. Proportion of participants with major osteoporotic fracture (hip, spine, wrist)
  2. Proportion of participants with any fracture
Long-term effects - health economic and labour market attachment, employment status | 5, 10 and 20 years after randomisation
  Employment status each participant
Long-term effects - health economic and labour market attachment, salary | 5, 10 and 20 years after randomisation
  Salary for each participant
Long-term effects - health economic and labour market attachment, absence | 5, 10 and 20 years after randomisation
  Number of absence days
Long-term effects - health economic and labour market attachment, sick leave | 5, 10 and 20 years after randomisation
  Proportion of participants with any sick leave
Long-term effects - health economic and labour market attachment, long-term sick leave | 5, 10 and 20 years after randomisation
  Proportion of participants with long-term sick leave (more than 4 weeks continuous sickness absence)

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, Ass. Prof., Study Chair — Department of Medicine, Copenhagen University Hospital - Amager and Hvidovre
Locations (10):
- Denmark (5):
  - The Department of Medicine and the Gastro Unit, Copenhagen University Hospital - Amager and Hvidovre, Copenhagen
  - Frederiksberg kommune: Social-, Sundheds- og Arbejdsmarkedsområdet, Frederiksberg
  - The Parker Institute, Copenhagen University Hospital - Bispebjerg and Frederiksberg, Frederiksberg
  - Hvidovre kommune: Center for Sundhed og Ældre, Hvidovre Sundhedscenter, Sundhed og Forebyggelse, Hvidovre
  - Gladsaxe kommune: Social- og Sundhedsforvaltningen, Sundhed og Rehabilitering, Søborg
- United Kingdom (5):
  - West Midlands RRDN, Birmingham
  - South West Peninsula RDN, Exeter, Exeter
  - Yorkshire and Humber RRDN (Leeds, Sheffield and Hull), Leeds
  - North West RRDN, Manchester
  - East of England RRDN, Norwich

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, the aim is to make a depersonalised dataset publicly available on e.g. ClinicalTrials.gov and/or the European Union (EU) Zenodo database (https://zenodo.org/). The final choice will reflect which platform(s) that are compliant with current legislation at that time
Supporting Information: Study Protocol, SAP
Time Frame: When the results have been published
Access Criteria: Researchers with a protocol for their planned study

REFERENCES:
- [Derived] Larsen SC, Heitmann BL, Wane S, Wielsoe S, Lindschou J, Jakobsen JC, Engstrom J, Specht IO, Christiansen AL, Jensen AKG, Bojsen-Moller KN, Bandholm T, Overbeck G, Kousgaard MB, Albury C, Reventlow S, Olsen KR, Kongstad LP, Madsbad S, Jebb SA, Dirksen C, Aveyard P, Waldorff FB; LightCOM team. Intensive weight loss intervention versus usual care in adults with obesity: a protocol for the LightCARE randomised clinical trial. BMJ Open. 2025 Oct 15;15(10):e107155. doi: 10.1136/bmjopen-2025-107155. PMID 41093354
- See also: LightCOM website — https://www.regionh.dk/lightcom/uk/Pages/default.aspx